CLINICAL TRIAL: NCT01233323
Title: Detection of Phrenic Nerve Stimulation Using Accelerometer and Electrogram Signals Study
Brief Title: Detection of Phrenic Nerve Stimulation Using Sensors' Signals
Acronym: DETECT PS
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: DETECT PS
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Heart Failure
Keywords: Phrenic nerve stimulation; Cardiac Resynchronization Therapy; Heart Failure; Heart Diseases
MeSH Terms: conditions — Heart Failure; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- All study patients (single arm study): All eligible patients will be included in the only study arm and will undergo study testing.

SUMMARY:
The purpose of this study is to collect sensor data from patients with implanted cardiac resynchronization devices who exhibit phrenic nerve stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Willing and capable of providing informed consent and of participating in all testing
* Age 18 or above or of legal age to give informed consent specific to national law
* Implanted with a Boston Scientific COGNIS™ family device
* Geographically stable and is available for follow-up procedures at a study centre

Exclusion Criteria:

* Patients that are pacemaker-dependent
* Women who are pregnant or plan to become pregnant during the study (method of assessment upon physician's discretion)
* Patients who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the patient is participating in a mandatory governmental registry
* Patients who are not expected to support approximately 30 minutes of study testing procedures
* Patients who are not mentally competent enough to provide feedback on PS during study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with a COGNIS™ CRT-D device
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Data collection | 3 months follow up
  Collect sensor data in patients with implanted CRT-D devices who exhibit phrenic nerve stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Glikson, MD, Principal Investigator — Heart Institute, Sheba Medical Center, Tel Hashomer, Israël
Locations (1):
- Deutsches Herzzentrum Berlin, Berlin, Germany